CLINICAL TRIAL: NCT05104541
Title: Impact of Weight Loss on Liver Fibrosis in Obese Patients With Cirrhosis
Brief Title: Impact of Weight Loss in Cirrhosis With Obesity and MAFLD
Acronym: WELCOME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-45
Record Dates: First submitted 2021-10-03; First posted 2021-11-03 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Liver Cirrhosis; Obesity
Keywords: Obesity; liver disease; nutrition; weight loss; fibrosis.
MeSH Terms: conditions — Liver Cirrhosis; Obesity; Liver Diseases; Weight Loss; Fibrosis

STUDY DESIGN:
Intervention Model Description: Prospective Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): In addition to standard pharmacological treatment this group would receive diet comprising of 20-25 kcal and 1.2gm protein per kg ideal body weight per day.
  The total distribution of the calories would be as 55-60% from carbohydrates, 25% from protein, and 20% from fat. The diet would be explained to the patient with the help of individual diet charts.
  Interventions: Other: Weight loss

INTERVENTIONS:
Other: Weight loss — In addition to standard pharmacological treatment this group would receive diet comprising of 20-25 kcal and 1.2gm protein per kg ideal body weight per day.
  The total distribution of the calories would be as 55-60% from carbohydrates, 25% from protein and 20% from fat. The diet would be explained to the patient with the help of individual diet charts.

SUMMARY:
Nutrition therapy is the cornerstone of medical therapy in patients with cirrhosis. 70% compensated patients with Chronic Liver Disease (CLD) are overweight or obese. Obesity in CLD augments decompensation, plausibly through increase in portal pressure. Moreover, the cardiometabolic risk factors are increased with increase in body weight, obesity also has an impact on the already compromised health-related quality of life of patients with CLD. Most feasible, safe, and widely used method of management of obesity is life-style modifications. Hypocaloric with normal to high protein diet along with moderate-intensity exercises have been practiced for weight reduction.

These kinds of dietary changes reduce body weight and may bring about favourable changes in the body composition (reduce the body fat percentage but at the same time preserving the lean body mass). Weight loss in obese patients with CLD would in turn improve the clinical outcome, reduce the hepatic complications, moreover weight loss may also improve health related quality of life, and other prognostic markers of the disease like fibroscan along with improvement in the associated metabolic derangements in patients with CLD. There is no Indian data in this context. Thus, through this trial, investigator would be able to ascertain an appropriate lifestyle-related non- intervention regimen that helps in the management of obesity in patients with cirrhosis. Not only that the baseline information of these obese patients with CLD would give us an idea or the profile of the body composition in terms of muscularity, adiposity, sarcopenic obesity (if any), of these patients with CLD.

DETAILED DESCRIPTION:
Liver disease is one of the main causes of hospital admissions worldwide and the 12th leading cause of mortality in many countries. Among all etiologies (toxic-metabolites, viral, autoimmune, and genetic disorders), nonalcoholic fatty liver disease (NAFLD) features as the most common cause, with increasing prevalence attributed to the epidemic of metabolic syndrome. According to the World Health Organization, in 2014, more than 30% of the United States population were obese and more than 60% overweight. Furthermore, 15% of all Western population and 35% of patients with obesity will develop steatohepatitis (NASH). Hence world over obesity is on a rise, the prevalence of obesity has consistently risen since past four decades in both genders. Indian similar scenario is seen not only in the urban but also in the rural population. This pandemic disease is attributed to both the increased amounts of processed foods high in fructose, sodium, and saturated fats, and the increasingly sedentary lifestyle. Obesity is considered a chronic state of low-grade inflammation, being associated with complications such as metabolic syndrome, type 2 diabetes, hypertension, and cardiovascular disease. It has also been linked with increased risks of certain cancers, such as colon, breast, breast, endometrium, kidney, esophagus, stomach, pancreas, and gallbladder. The combination of obesity, insulin resistance, and NASH is also thought to increase the risk of Hepatocellular Carcinoma (HCC). Most of all obesity in cirrhotics accelerates decompensation plausibly through an increase in portal hypertension. The risk of first clinical decompensation of cirrhosis is approximately three times higher in obese cirrhotics compared to those with normal weight. There are innumerable randomized controlled trials examining the role of various kinds of weight-loss diets and regimens in NAFLD patients, namely Mediterranean diets, Ornish diets, south beach diets, Atkins diets, Zone diet, weight watcher's diets, etc. However, once cirrhosis sets in or is diagnosed the concept of malnutrition akin to undernutrition is the prime consideration in a patient which baffles the physicians. The nutritional guidelines either European Society of Parenteral and Enteral Nutrition (ESPEN) or American Society of Parenteral and Enteral Nutrition (ASPEN) have always focused on a high calorie and a high protein diet in cirrhosis. These guidelines have not even touched upon the topic of obesity in cirrhosis. Moreover, for decades, investigator have been obsessed with the idea of protein restriction in patients with cirrhosis. In the recent past, our attention is drawn towards the other end of the spectrum of malnutrition i.e. obesity, which has been steadily on the rise world over and cirrhotics are no exception. Obesity is associated with poor survival, severe hepatic decompensation, poor post-transplantation outcomes as well as greater difficulty in liver transplantation, and also higher non-response to antiviral therapy in patients with cirrhosis. Hence weight reduction is the standard of care in such patients. A few studies have examined the role of a monitored exercise program including resistance training including cycle ergometric exercises have been shown to favorably change the body composition but none have been done in obese cirrhotics with the aim of weight loss. At the same time, low-calorie and even very-low-calorie ketogenic diets have been tried in obese cirrhosis and published as case series. Based on the magnitude of the problem of obesity in CLD and its detrimental impact on the clinical outcome investigator propose to assess the impact of weight loss with low calorie, high protein diet and moderate physical activity (lifestyle modifications- a non-pharmacological strategy) on liver fibrosis, body composition changes, functional capacity, clinical outcome in obese cirrhotics in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18 and 65 years.
* Obese cirrhotics of any etiology.
* BMI > 30

Exclusion Criteria:

* Patients with oChild B (8,9) and C oMELD>20

  * High-risk varices
  * HPS/ pleural effusion
  * Alcoholic Hepatitis
  * Chronic Kidney Disease, cardiac, neurological diseases
  * HCC
  * Pregnancy
  * Unwilling patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-11-09 (Estimated); Study Completion 2023-11-09 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with change in liver fibrosis with 10% weight loss in 3 months in an obese patient with CLD. | 3 months

SECONDARY OUTCOMES:
Effect of weight loss (10%) in three months on Insulin resistance (HOMA- IR) | 3 months
  Insulin resistance will be measured at baseline and at 3 months
Effect of weight loss (10%) in three months on Triglyceride levels | 3 months
  Triglyceride levels will be measured at baseline and at 3 months
Effect of weight loss (10%) in three months on blood sugar levels as a component of metabolic syndrome | 3 months
  Blood sugar levels will be noted at baseline and at 3 months
Effect of weight loss (10%) in three months on central obesity as a component of metabolic syndrome | 3 months
  Central obesity will be noted at baseline and at 3 months
Effect of weight loss (10%) in three months on high density lipoprotein (HDL) as a component of metabolic syndrome | 3 months
  High density lipoprotein (HDL)metabolic syndrome will be noted at baseline and at 3 months
Effect of weight loss (10%) in three months on metabolic syndrome | 3 months
  Components of metabolic syndrome will be noted at baseline and at 3 months
Effect of weight loss (10%) in three months on body composition- bio electrical impedance | 3 months
  Body composition by bioelectrical impedance will be measured at baseline and at the end of three months
Effect of weight loss (10%) in three months on anthropometric mid arm muscle circumference (MAMC) | 3 months
  Mid amr muscle circumference (MAMC) will be measured at baseline and at the end of three months
Effect of weight loss (10%) in three months on anthropometric Mid upper arm circumference (MUAC) | 3 months
  Mid upper arm circumference (MUAC) will be measured at baseline and at the end of three months
Effect of weight loss (10%) in three months on anthropocentric tricep fold thickness (TSF) | 3 months
  Tricep fold thickness (TSF) will be measured at baseline and at the end of three months
Effect of weight loss (10%) in three months on functional capacity | 3 months
  Functional capacity will be measured by hand grip dyanamometer at baseline and at the end of three months
Effect of weight loss (10%) in three months on Pro inflammatory marker- (Tumor Necrosis Factor) TNF-alpha | 3 months
  Pro inflammatory marker will be noted at baseline and at 3 months
Effect of weight loss (10%) in three months on Pro inflammatory marker -IL-6 | 3 months
  Pro inflammatory marker will be noted at baseline and at 3 months
Effect of weight loss (10%) in three months on Anti inflammatory marker -Adiponectin | 3 months
  Anti inflammatory marker (Adiponectin) will be noted at baseline and at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shiv Kumar Sarin, MD, DM, FNA, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided